CLINICAL TRIAL: NCT05473299
Title: Prospective, Non-randomized Pivotal Clinical Study to Assess the Safety and Performance of the Xeltis Hemodialysis Access Graft: aXess Pivotal Study
Brief Title: Xeltis Hemodialysis Access Graft: aXess Pivotal Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xeltis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XEL-CR-10
Record Dates: First submitted 2022-07-06; First posted 2022-07-25 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: End-stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- aXess graft (Experimental)
  Interventions: Device: Xeltis Hemodialysis Access (aXess) graft

INTERVENTIONS:
Device: Xeltis Hemodialysis Access (aXess) graft — The aXess graft is a sterile, regenerative biodegradable polymer-based vascular graft, consisting of a tubular structure with a 6mm inner diameter. It is comprised of a highly porous polymer matrix and an embedded electropolished nitinol reinforcement layer (Strain Relief System). The aXess graft is able to support both straight and loop configurations and may be implanted in the upper arm and forearm.

SUMMARY:
A prospective, single arm, non-randomized pivotal study to evaluate the safety and performance of the Xeltis hemodialysis access graft in subjects older than 18 years with end-stage renal disease, who plan to undergo hemodialysis for at least the first 6 months after study access creation.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with end-stage renal disease (ESRD) who require placement of an AVG in the upper extremity to start or maintain hemodialysis therapy
2. At least 18 years of age at screening
3. Suitable anatomy (e.g. a target vein with a minimum diameter of 5mm) for the implantation of an aXess graft
4. The patient, or legal representative, has been informed about the nature of the study, agrees to its provisions, and has provided written informed consent
5. The patient has been informed and agrees to pre- and post- procedure follow-up
6. Life expectancy of at least 12 months

Exclusion Criteria:

1. History or evidence of severe cardiac disease (NYHA Functional Class IV and/or EF <25%), myocardial infarction within six months of study enrolment, ventricular tachyarrhythmias requiring continuing treatment, or unstable angina
2. Uncontrolled or poorly controlled diabetes
3. Abnormal blood values that could influence patient recovery and or/ graft hemostasis
4. Reduced liver function, defined as: >2x the upper limit of normal for serum bilirubin, International Normalized Ratio (INR) >1.5 or prothrombin time (PT) >18 seconds
5. Any active local or systemic infection
6. Known heparin-induced thrombocytopenia
7. Known active bleeding disorder and/or any coagulopathy or thromboembolic disease
8. Allergies to study device (nitinol) or agents/medication, such as contrast agents or aspirin, that can't be controlled medically
9. Anticipated renal transplant within 6 months
10. Known or suspected central vein obstruction on the side of planned graft implantation
11. Previous dialysis access graft in the operative limb unless the aXess graft can be placed more proximally than the previous failed graft
12. Previous enrolment in this study
13. Subject is participating in another study
14. Pregnant or breastfeeding woman or woman in fertile period not taking adequate contraceptives
15. Any other condition which, in the judgement of the investigator would preclude adequate evaluation for the safety and performance of the study conduit

Intra-operative exclusion criteria:

1. Unsuitable anatomy to implant the aXess graft (e.g. target vein and/or artery diameter smaller than anticipated; severe calcification)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-11-04 (Actual); Primary Completion 2025-06-23 (Actual); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary patency rate | 6 months
  Defined as the interval between vascular access creation and the first intervention to maintain or restore patency.
Freedom from device-related SAE during the first 6 months | up to 6 months

SECONDARY OUTCOMES:
Implantation success rate | 1 day, from moment of implant until end of procedure day
  Defined as a technically successful aXess graft implantation in the planned configuration, free from kinking and tension in the anastomoses. This is assessed at the procedure day itself.
Patency (primary, primary assisted, secondary, and functional) rates | 6, 12, 18, 24 and 60 months
  Primary patency: Defined as the interval between vascular access creation and the first intervention to maintain or restore patency.
  Assisted primary patency: Defined as the interval between vascular access creation and the first occlusion (thrombosis), including interventions (operative or endovascular) aimed to maintain the functionality the vascular access.
  Secondary patency: Defined as the interval between vascular access creation and abandonment with or without interventions (operative or endovascular) aimed to maintain the functionality the vascular access, including occurrence of a censored event (death, change of modality, loss of follow-up).
  Functional patency: Defined as the interval between first cannulation and abandonment, including occurrence of a censored event (death, change of modality, loss of follow-up).
Time (expressed in months) to first intervention and to access abandonment | 60 months
Rate of access-related interventions required to achieve/maintain patency | 6, 12, 18, 24, and 60 months
Freedom from device-related SAE | 12, 18, 24, and 60 months
Rate of access site infections | 6, 12, 18, 24, and 60 months
Proportion of hemodialysis sessions completed via central venous catheter (CVC) during the first 12 months of access creation and access cannulation, irrespective of access abandonment | 12 months
Time to first cannulation | 12 months
Following first cannulation, number of days with CVC in situ (catheter contact time) during the first 12 months, irrespective of access abandonment | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Gargiulo, Prof, Principal Investigator — Policlinico di Sant'Orsola; An de Vriese, Dr, Principal Investigator — AZ Sint-Jan AV
Locations (22):
- Belgium (3):
  - AZ Sint Jan Brugge, Bruges
  - ZOL Genk, Genk
  - UZ Ghent, Ghent
- Universitätsklinikum Köln, Cologne, Germany
- Greece (2):
  - LAIKO General Hospital of Athens, Athens
  - University General Hospital of Patras, Pátrai
- Italy (5):
  - Ospedali Riuniti Torrette di Ancona, Ancona
  - Policlinico di Bari, Bari
  - Policlinico di Sant'Orsola, Bologna
  - Università degli studi di Padova / Azienda ospedaliera di Padova, Padua
  - Universita degli studi dell'Insubria, Varese
- Pauls Stradins Clinical University Hospital, Riga, Latvia
- Poland (2):
  - Private hospital MedPolonia Poznan, Poznan
  - The Lower Silesia Center of Heart Diseases MEDINET, Wroclaw
- Portugal (3):
  - Santa Maria Hospital, Lisbon
  - Grupo de Estudos Vasculares, Porto
  - DaVita Sacavém, Sacavém
- Spain (3):
  - Bellvitge University Hospital, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitario de la Ribera, Valencia
- United Kingdom (2):
  - University Hospitals Birmingham - QE, Birmingham
  - Queen Elizabeth University Hospital, Glasgow

IPD SHARING:
Plan to Share IPD: No